CLINICAL TRIAL: NCT05059210
Title: Primary Care Implementation and Evaluation of Coach McLungs, an Asthma Shared Decision-making Intervention, Across a Large Healthcare System
Brief Title: Primary Care Implementation and Evaluation of Coach McLungs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00082608; 1R01HL151854-01A1 (NIH)
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Asthma
Keywords: Asthma; Shared Decision Making
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Pragmatic, stepped-wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Coach McLungs not yet implemented in practice
- Intervention (Active Comparator): Coach McLungs Implemented in Practice
  Interventions: Behavioral: Coach McLungs Intervention

INTERVENTIONS:
Behavioral: Coach McLungs Intervention — Practices have received implementation of Coach McLungs
  Arms: Intervention

SUMMARY:
The goal of this study is to evaluate the implementation of the Coach McLungsSM shared decision making (SDM) intervention into primary care across a large healthcare system. Coach McLungsSM is a virtual evidence-based asthma intervention with built-in asthma education and clinical decision support. All asthma patients aged 5-17 who attend these practices will be assessed for uncontrolled asthma. Asthma exacerbations attributed to emergency department visits, hospitalizations, and oral steroid use, will be evaluated to serve as surrogate measures for patient-centered asthma outcomes.

DETAILED DESCRIPTION:
Changing behavior of health providers can be challenging, and significant gaps exist in our knowledge of how to best implement new medical evidence into everyday practice. Numerous individual- and system-level factors contribute to poor asthma outcomes which persist due to the lack of a comprehensive approach for asthma care that is scalable, sustainable, and widely disseminated. Improved asthma outcomes are associated with effective communication strategies between the patient and provider. Shared decision making (SDM) is a patient-centered process in which patients and providers work together to make decisions and select tests, treatments, and care plans based on evidence that balances risks with patient preferences and values. Previous studies, including a PCORI-funded dissemination study, have shown that SDM is associated with improved outcomes for asthma patients in primary care. The implementation of Coach McLungsSM, a virtual evidence-based asthma SDM intervention with built-in asthma education and clinical decision support, will be evaluated as it is implemented into primary care practices across a large healthcare system. Atrium Health, the 2nd largest virtually integrated healthcare system in the nation, with over 14 million patient visits per year and the region's largest primary care network, provides an ideal venue to evaluate implementation into primary care. Coach McLungsSM will be fully integrated into the electronic medical record at all primary care practices. All asthma patients aged 5-17 who attend these practices will be assessed for uncontrolled asthma. The goal of this study will be to evaluate the implementation of the Coach McLungsSM SDM intervention into primary care. Implementation will be guided using the Expert Recommendations for Implementing Change (ERIC), a compilation of implementation strategies, and evaluated using the RE-AIM (Reach Effectiveness, Adoption, Implementation, Maintenance) framework. Research questions are: How best can Coach McLungsSM SDM asthma intervention be implemented into primary care? Will use of Coach McLungsSM in primary care improve outcomes for patients with uncontrolled asthma? After convening a Stakeholder Advisory Committee (SAC) composed of providers, researchers, patients, stakeholders with expertise in implementation science, asthma research and advocacy, the Coach McLungsSM SDM intervention will be implemented into primary care practices using a stepped wedge randomized control study design. Providers and staff will be trained in SDM communication and use of the Coach McLungsSM tool. Changes in emergency department visits, hospitalizations, and oral steroid use, which serve as surrogate measures for patient-centered asthma outcomes will be evaluated. The SAC will use an iterative process improvement method and give best practice recommendations back to the practices for implementation improvement. Findings will be disseminated through local stakeholders, practice-based research networks, asthma advocacy national organizations, and academic research meetings for healthcare, primary care, and asthma.

ELIGIBILITY:
Inclusion Criteria:

* Established mild, moderate, or severe persistent asthma
* English or Spanish speaking.

Exclusion Criteria:

• Decisional impaired or mentally incompetent

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Asthma Exacerbations | 6 Months
  Participant utilization data of ED visits and hospitalizations for asthma exacerbations will be extracted from the electronic data warehouse (EDW) for participants who have a diagnosis of asthma (ICD-10 code J45.XXX) irrespective of intervention, allowing measurement of any outcome improvements over the life of the study.

SECONDARY OUTCOMES:
Number of Participants with Asthma Exacerbations | 12 months
  Participant utilization data of ED visits and hospitalizations for asthma exacerbations will be extracted from the electronic data warehouse (EDW) for participants who have a diagnosis of asthma (ICD-10 code J45.XXX) irrespective of intervention, allowing measurement of any outcome improvements over the life of the study.
Number of Participants with Asthma Exacerbations | 18 months
  Participant utilization data of ED visits and hospitalizations for asthma exacerbations will be extracted from the electronic data warehouse (EDW) for participants who have a diagnosis of asthma (ICD-10 code J45.XXX) irrespective of intervention, allowing measurement of any outcome improvements over the life of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Tapp, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ludden T, O'Hare K, Shade L, Reeves K, Patterson CG, Tapp H. Implementation of Coach McLungsSM into primary care using a cluster randomized stepped wedge trial design. BMC Med Inform Decis Mak. 2022 Nov 4;22(1):285. doi: 10.1186/s12911-022-02030-1. PMID 36333727